CLINICAL TRIAL: NCT05512338
Title: Patient Motivation and Adherence to Rehabilitation Exercise Recommendations in Patients With Chronic Low Back Pain- PACT vs. Usual Physiotherapy
Brief Title: Motivation and Adherence to Exercise Recommendations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ladislav Batalik, Ladislav Batalik, PT, PhD, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHO/G5
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACT treatment group (Experimental): PACT treatment will include an initial physical assesment with feedback, identification of value-based goals, individualized physical exercise based on the DNS concept, manual therapy, addressing barriers and facilitators to self-management, and skills training to promote psychological flexibility.
  Interventions: Other: Treatment
- Usual physiotherapy care group (Active Comparator): UC will include an initial physical assesment with feedback, treatment considered suitable by their treating physiotherapist that will be based on exercises according to the DNS concept and manual therapy.
  Interventions: Other: Active control group

INTERVENTIONS:
Other: Treatment — ACT-informed interventions combined with standard physiotherapy methods.
  Arms: PACT treatment group
Other: Active control group — Standard physiotherapy methods.
  Arms: Usual physiotherapy care group

SUMMARY:
Low back pain is a common condition that occurs in up to 70% of the population in industrialized countries and is the second most common cause of work inability. Physiotherapy is the usual treatment for low back pain. Recent studies showed that combining theory-based psychological methods with physiotherapy can enhance the effectiveness of physiotherapy treatment for people with chronic low back pain.

One promising approach to treating chronic pain is PACT - Physiotherapy informed by Acceptance and Commitment Therapy (ACT), a form of cognitive-behavioral therapy. PACT aims to increase psychological flexibility and focus on improving function rather than reducing pain.

According to several studies, the effects of ACT can be maintained up to 3 years post-treatment, which is essential in a condition such as chronic pain and its typical relapses.

According to self-determination theory (SDT), facilitating an environment of acceptance and autonomy support enhances treatment motivation, thus offering a good interface for applying SDT´s research concepts to ACT interventions.

The primary objective of this study is to investigate the impact of physiotherapists´ autonomy-supportive behavior within PACT on the motivation process in chronic low back pain patients. Other objectives are to evaluate the efficacy of PACT on the functioning and disability due to CLBP, adherence to recommended physical activity, and the acceptance of pain.

This prospective, randomized controlled trial will include 2 treatment groups (PACT treatment group and Usual physiotherapy Care group[UC]) in 1:1 ratio. Participants in the PACT treatment group will undergo a physiotherapy intervention guided by ACT principles.

Participants randomized to UC will receive treatment considered suitable by their treating physiotherapist, including exercises based on the DNS concept and manual therapy.

Regardless of group assignment, all participants will undergo 6 physiotherapy face-to-face interventions lasting 45 minutes, each once a week.

Study outcomes will include measures of treatment motivation, perceived degree of autonomy support within the care settings, functioning, and disability, adherence to recommended physical activity, and acceptance of pain.

While we acknowledge the value of usual physiotherapy care, CLBP is best suited to a biopsychosocial model for care. Further research is needed to understand which underlying processes and components are causing the improvement.

DETAILED DESCRIPTION:
Eligible participants will be randomly assigned to one of the treatment groups. All subjects will undergo 6 weeks of weekly face-to-face sessions.

PACT treatment will include an initial physical assesment with feedback, identification of value-based goals, individualized physical exercise based on the DNS concept, manual therapy, addressing barriers and facilitators to self-management, and skills training to promote psychological flexibility.

UC will include an initial physical assesment with feedback, treatment considered suitable by their treating physiotherapist that will be based on exercises according to the DNS concept and manual therapy.

The self-report questionnaires will be completed by participants at baseline and 6 weeks, all to be completed at home.

Treatment will be provided by an experienced physiotherapist and will be conducted in a private room.

To avoid contamination, the same clinician will deliver both PACT and UC as CBT-based methods are sometimes employed within usual physiotherapy care.

A clinical psychologist and expert in the ACT will provide training. There will be group face-to-face training that will last 2 days followed by self-experience group training that will last 6 weeks (2 hours/week).

All PACT sessions will be audio-recorded to assesing treatment fidelity. Recordings will be used for supervision. Supervisor will be a clinical psychologist experienced in ACT and will review one tape per month.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 18
* Chronic low-back pain longer than 12 weeks
* Scoring more than 3 points in Roland-Morris Disability Questionnaire (RMDQ)
* Adequate understanding of spoken and written czech language

Exclusion Criteria:

* Prior treatment from cognitive-behavioural therapy pain management at any time and other physiotherapy treatment in the previous 6 months
* Injection therapy within 3 months
* Specific medically diagnosed lubar spine pathology (eg, fracture, cancer)
* Deteorating neurological sings
* Patients with current psychiatric illness
* Current alcohol or drug misuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Treatment motivation | Change from baseline to 6 weeks
  We will assess individual differences in the types of motivation to exercise by using Exercise Self-Regulation Questionnaire. Values ranges from 1-7, higher scores mean a better outcome.

SECONDARY OUTCOMES:
Autonomy support from from physiotherapist | Change from baseline to 6 weeks
  We will assess patients´ perception of their physiotherapist autonomy support using Health Care Climate Questionnaire. Values ranges from 1-7, higher scores mean a better outcome.
Adherence to recommended physical activity | Change from baseline to 6 weeks
  Adherence to prescribed home exercise will be obtained by Exercise Adherence Rating Scale questionnaire.Values ranges from 1-5, lower scores mean a better outcome.
Functioning and disability | Change from baseline to 6 weeks
  Patient functioning and diability will be measured by the Roland-Morris Disability Questionnaire. Values ranges from 0-24, lower scores mean a better outcome.
Acceptance of Pain | Change from baseline to 6 weeks
  Acceptance of Pain will be measured by the Chronic Pain Acceptance Questionnaire-8. Values ranges from 0-6, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Marketa Nevelikova, PT, Study Director — Department of Rehabilitation, University Hospital Brno, Czech Republic
Locations (1):
- University Hospital Brno, Brno, Czechia

REFERENCES:
- [Derived] Nevelikova M, Zlamal F, Dosbaba F, Su JJ, Batalik L. Motivation to exercise in patients with chronic low back pain. BMC Musculoskelet Disord. 2025 Mar 6;26(1):226. doi: 10.1186/s12891-025-08461-x. PMID 40050856